CLINICAL TRIAL: NCT03414489
Title: Expanded Access to ABC-108, A Phase IIA Study of ABC294640 in the Treatment of Patients With Advanced,Unresectable Intra-hepatic, Perihilar and Extra-Hepatic Cholangiocarcinoma
Brief Title: Expanded Access for the Treatment of Advanced Cholangiocarcinoma With ABC294640 (Yeliva ®)
Status: No longer available | Type: Expanded Access
Sponsor: RedHill Biopharma Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: ABC-108-EA
Record Dates: First submitted 2018-01-22; First posted 2018-01-30 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Cholangiocarcinoma; Cholangiocarcinoma Non-resectable; Cholangiocarcinoma, Perihilar; Cholangiocarcinoma, Extrahepatic; Cholangiocarcinoma, Intrahepatic
Keywords: Clinical Trial, Phase II; Multicenter Trials; Clinical Study; Clinical Trials, Non-Randomized; Oral capsule; Single arm; Anti-cancer; Anti-inflammatory; ABC294640; Expanded Access Program; Compassionate Use; Special Access Program; Yeliva ®; opaganib
MeSH Terms: conditions — Cholangiocarcinoma; Klatskin Tumor | interventions — 3-(4-chlorophenyl)-adamantane-1-carboxylic acid (pyridin-4-ylmethyl)amide

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: ABC294640

SUMMARY:
This is an expanded access program (EAP) for eligible participants who do not qualify for participation in, or who are otherwise unable to access, the ongoing clinical trial ABC-108. This program is designed to provide access to ABC294640 (Yeliva ®) for treatment of cholangiocarcinoma (CCA) prior to approval by the local regulatory agency. Availability will depend on territory eligibility. Participating sites will be added as they apply for and are approved for the EAP. An oncologist must decide whether the potential benefit outweighs the risk of receiving an investigational therapy based on the individual patient's medical history and program eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of cholangiocarcinoma
2. Ineligible to participate in the ABC294640 clinical trial for the treatment of cholangiocarcinoma or geographically inaccessible to the trial.
3. Judged by the treating oncologist to be medically suitable for treatment with ABC294640
4. Willing and able to provide written, signed informed consent
5. Approval by RedHill of the treating oncologist's clinical trial experience for the purpose of making ABC294640 available
6. Regulatory approval by the appropriate jurisdiction

Exclusion Criteria:

1. Any medical condition that may cause treatment with ABC294640 to be potentially harmful as judged by RedHill

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

REFERENCES:
- [Background] Ding X, Chaiteerakij R, Moser CD, Shaleh H, Boakye J, Chen G, Ndzengue A, Li Y, Zhou Y, Huang S, Sinicrope FA, Zou X, Thomas MB, Smith CD, Roberts LR. Antitumor effect of the novel sphingosine kinase 2 inhibitor ABC294640 is enhanced by inhibition of autophagy and by sorafenib in human cholangiocarcinoma cells. Oncotarget. 2016 Apr 12;7(15):20080-92. doi: 10.18632/oncotarget.7914. PMID 26956050
- [Background] Beljanski V, Knaak C, Smith CD. A novel sphingosine kinase inhibitor induces autophagy in tumor cells. J Pharmacol Exp Ther. 2010 May;333(2):454-64. doi: 10.1124/jpet.109.163337. Epub 2010 Feb 23. PMID 20179157
- [Background] French KJ, Zhuang Y, Maines LW, Gao P, Wang W, Beljanski V, Upson JJ, Green CL, Keller SN, Smith CD. Pharmacology and antitumor activity of ABC294640, a selective inhibitor of sphingosine kinase-2. J Pharmacol Exp Ther. 2010 Apr;333(1):129-39. doi: 10.1124/jpet.109.163444. Epub 2010 Jan 8. PMID 20061445
- [Result] Britten CD, Garrett-Mayer E, Chin SH, Shirai K, Ogretmen B, Bentz TA, Brisendine A, Anderton K, Cusack SL, Maines LW, Zhuang Y, Smith CD, Thomas MB. A Phase I Study of ABC294640, a First-in-Class Sphingosine Kinase-2 Inhibitor, in Patients with Advanced Solid Tumors. Clin Cancer Res. 2017 Aug 15;23(16):4642-4650. doi: 10.1158/1078-0432.CCR-16-2363. Epub 2017 Apr 18. PMID 28420720